CLINICAL TRIAL: NCT06878352
Title: Impact of Educational Intervention Protocol on the Level of Knowledge, Clinical Control and Lung Function of People With Asthma: Randomized Controlled Clinical Trial
Brief Title: Impact of Educational Intervention Protocol on the Level of Knowledge, Clinical Control and Lung Function of People With Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Renata Ramos Tomaz Barbosa, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6.968.418
Record Dates: First submitted 2025-02-19; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Asthma
Keywords: Asthma; Heath Education; Spirometry; Respiratory Tract Disease
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher responsible for the baseline and endpoint assessments will be blinded to the participant's group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): The control group will receive standard follow-up according to the clinic routine.
- Educational intervention BUNDLE (Experimental): The experimental group will undergo an educational intervention BUNDLE, prepared in accordance with the recommendations of the Global Initiative for Asthma- GINA (2024), and will cover topics on the etiopathogenesis and pathophysiology of asthma, inhaler treatment, precipitating factors for crises, self-management skills, environmental control, as well as the importance of drawing up a written therapeutic plan and regular medical follow-up.
  Interventions: Other: Educational intervention BUNDLE, prepared in accordance with the recommendations of the Global Initiative for Asthma- GINA (2024)).

INTERVENTIONS:
Other: Educational intervention BUNDLE, prepared in accordance with the recommendations of the Global Initiative for Asthma- GINA (2024)). — The educational intervention bundle was designed in accordance with the recommendations of GINA (2024), and will cover topics on the etiopathogenesis and pathophysiology of asthma, inhaler treatment, precipitating factors for crises, self-management skills, environmental control, as well as the importance of drawing up a written therapeutic plan and regular medical follow-up.
  The educational intervention will be offered as a group activity and will be conducted in a single meeting, lasting approximately sixty minutes. Users will attend a standardized dialogical lecture using audiovisual resources, where they will have the opportunity to discuss and answer any questions related to the topics covered. At the end of the intervention, participants will receive a booklet containing all the points covered in the intervention, as well as a diary to record the amount of medication used, visits to the emergency room and asthma-related hospitalizations.
  Other Names: Health Education; Educational Intervention; Bundle
  Arms: Educational intervention BUNDLE

SUMMARY:
The goal of this randomized controlled clinical trial is to evaluate the effects of a proposed educational intervention on people with asthma. The main question it aims to contribute to a better understanding of the effectiveness of educational intervention strategies in people with asthma.

Participants allocated to the control group will receive standard follow-up according to the clinic routine. Participants allocated to the experimental group will undergo an educational intervention BUNDLE, prepared in accordance with the recommendations of the Global Initiative for Asthma- GINA (2024).

DETAILED DESCRIPTION:
People with asthma will participate in the study, from the Pulmonary Function Clinic of the Department of Physiotherapy at Federal University of Paraíba - UFPB. Spirometry data, knowledge about asthma and correct control over inhalation therapy, clinical control of the disease using the Asthma Control Test (ACT) and C-ACT questionnaire, number of asthma attacks, amount of medication used, hospitalizations and visit to the emergency room in the last 4 weeks will be assessed. Assessments will be carried out at the first contact (baseline) and twelve weeks after the first contact.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Assisted by the Pulmonary Function Clinic
* Ventilatory dysfunction assessed by spirometry

Exclusion Criteria:

* Obesity
* Treatment with systemic corticosteroids
* Previous chest surgery
* Unable to perform any of the proposed assessment steps

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
clinical asthma control | Baseline and 4 weeks
  Asthma Control Test (ACT)/Childhood Asthma Control Test (C-ACT) score. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Retention of information about asthma knowledge and inhalation therapy | Baseline and 4 weeks
  Number of correct answers obtained from the asthma knowledge questionnaire at the end of the educational intervention

SECONDARY OUTCOMES:
hospitalizations and emergency room visits | Baseline and 4 weeks
  number of hospitalizations and emergency room visits in the last four months
Pulmonary function - Spirometry | Baseline and 4 weeks
  Predicted percentages of spirometric variables such as the values of Forced Expiratory Volume in 1 second (FEV1) and Forced Vital Capacity (FVC) because the correlation between these values can indicate the presence of respiratory disorders such as asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Function Clinic of the Department of Physiotherapy at Federal University of Paraiba, João Pessoa, Paraíba, Brazil

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT06878352/Prot_SAP_ICF_000.pdf